CLINICAL TRIAL: NCT02828254
Title: A Follow-up Evaluation Study of the Safety and Efficacy of PRI-724 Administration in Patients With Cirrhosis Due to Hepatitis C
Brief Title: A Follow-up Evaluation Study of PRI-724-1101
Status: Completed | Type: Observational
Sponsor: Komagome Hospital (Other)
Collaborators: Prism Pharma Co., Ltd. (Industry); Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Principal Investigator, Kiminori Kimura, MD, MD, Komagome Hospital
Other Study IDs: PRI-724-1102; UMIN000014891 (Other: UMIN (University Hospital Medical Information) CTR)
Record Dates: First submitted 2016-06-15; First posted 2016-07-11 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis C Virus-infected Cirrhosis
MeSH Terms: interventions — ICG 001

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PRI-724
  Other Names: CBP-beta-catennin inhibitor; OP-724

SUMMARY:
The purpose of this study To evaluate the safety and efficacy of PRI-724 administration in patients with cirrhosis due to hepatitis C by 12-month follow-up.

DETAILED DESCRIPTION:
This is a single-center, nonintervention, open-label, observational study in subjects who received the study drug (identification code: PRI-724) in Study 1101 to follow up the safety and disease condition of cirrhosis after administration for 12 months.

In Study 1101, one cycle consisted of 2 weeks with one-week continuous i.v. administration of PRI-724 followed by a one-week observation period. Treatment with a total of six cycles (duration of treatment, 12 weeks) was performed.

In this study, the subjects in each cohort in Study 1101 (PRI-724 dose: Cohort 1, 10 mg/m2/day; Cohort 2, 40 mg/m2/day; Cohort 3, 160 mg/m2/day) were followed up and observed for 12 months after administration.

In Study 1101, target number of subjects was 6 subjects in each cohort, a total of 18 subjects. However, the number of registered subjects was 7 subjects in Cohort 1, 7 subjects in Cohort 2, and 2 subjects in Cohort 3, a total of 16 subjects. Safety analysis set was 6 subjects, 6 subjects, and 2 subjects, respectively, a total of 14 subjects. Target number of the subjects in this study was the same as that in Study 1101; however, of the subjects in Study 1101, 5 subjects in Cohort 1 and 3 subjects in Cohort 2 consented to participate in this study (Study 1102).

ELIGIBILITY:
Inclusion Criteria:

1. Having been administered PRI-724 in Study 1101 after being confirmed to meet the inclusion criteria and not to meet the exclusion criteria and consenting to participate in the study.
2. Having provided voluntary written consent for participation in this study.

Exclusion Criteria:

1. Patients who are pregnant or may be pregnant, or who desire to become pregnant or may be pregnant during the clinical study [excluding patients who have undergone a sterilization procedure or postmenopausal patients (if amenorrhea without medical reasons continues more than 12 months), patients who are nursing.
2. Patients who do not consent to practice birth control during the clinical study (including male patients).
3. Patients with serious allergy to contrast media or a history thereof.
4. Patients with a history of drug or alcohol addiction within five years at the time of providing written consent or a history of drug or alcohol abuse within the past one year.
5. Patients contraindicated for liver biopsy. However, this criterion will not apply to a patient who has turned out to be contraindicated for liver biopsy after having been administered PRI-724 in Study 1101.
6. Patients who participated in another clinical trial, except PRI-724-1101 trial, within 30 days at the time of providing written consent.
7. Patients who have discontinued administration of PRI-724 in Study 1101 due to death or other reasons and become lost for follow-up.
8. Other, at the point when Study 1101 has been completed (or discontinued), patients who are judged inappropriate for inclusion in the study by the investigator for such reasons as the presence of serious pathological condition.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PRI-724 administration in patients with cirrhosis due to hepatitis C
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Safety: Incidences of adverse events and adverse drug reactions | 12 months after completion of the clinical trial, PRI-724-1101
  The data will be aggregated by each adverse events, cohort and Child-Pugh score

SECONDARY OUTCOMES:
Incidence of liver cancer | 12 months after completion of the clinical trial, PRI-724-1101
  The data will be aggregated by each cohort and Child-Pugh score
Child-Pugh Score | 12 months after completion of the clinical trial, PRI-724-1101
  The data will be aggregated by each cohort and Child-Pugh score
Liver biopsy (Only in applicable patients) | 12 months after completion of the clinical trial, PRI-724-1101
  The data will be aggregated by each cohort and Child-Pugh score
Serum albumin level | 12 months after completion of the clinical trial, PRI-724-1101
  The data will be aggregated by each cohort and Child-Pugh score
Serum fibrosis marker level(s) | 12 months after completion of the clinical trial, PRI-724-1101
  The data will be aggregated by each cohort and Child-Pugh score
Ascitic fluid level | 12 months after completion of the clinical trial, PRI-724-1101
  The data will be aggregated by each cohort and Child-Pugh score
Improvement rate of lower leg edema | 12 months after completion of the clinical trial, PRI-724-1101
  The data will be aggregated by each cohort and Child-Pugh score

CONTACTS AND LOCATIONS:
Overall Officials: Kiminori Kimura, MD, Principal Investigator — Komagome Metropolitan Hospital
Locations (1):
- Tokyo metropolitan Komagome Hospital, Tokyo, Japan